CLINICAL TRIAL: NCT00495066
Title: A Multicenter Treatment Protocol for Expanded Access Use of Ipilimumab (BMS-734016) Monotherapy in Subjects With Unresectable Stage III or Stage IV Melanoma
Brief Title: Compassionate Use Trial for Unresectable Melanoma With Ipilimumab
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA184-045
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Intravenous Solution, Intravenous, Ipilimumab 3 mg/kg, Ipilimumab - one dose every 3 wks for a total of 4 doses. Subjects who are eligible may receive another 4 doses given every 3 wks; Until disease progression, unacceptable toxicity or withdrawal of consent

SUMMARY:
The primary objective of the study is to provide treatment with Ipilimumab to subjects who have serious or immediately life-threatening unresectable Stage III or Stage IV melanoma, who have no alternative treatment options, and whose physicians believe, based upon available data on benefit and risk, that it is appropriate to administer Ipilimumab at a dose of 3 mg/kg induction (with re-induction, if eligible), or for eligible subjects previously enrolled in Ipilimumab studies CA184-042, CA184-078, CA184-087, MDX010-16, or MDX010-20.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Histologically confirmed Stage III (unresectable) or Stage IV melanoma
* Must have failed at least one systemic therapy for malignant melanoma or be intolerant to at least one prior systemic treatment. Note: Enrollees must not be eligible for a clinical study with Ipilimumab
* Subjects with asymptomatic brain metastases are eligible
* Primary ocular and mucosal melanomas are allowed
* Must be at least 28 days since treatment with chemotherapy, biochemotherapy, or immunotherapy, and recovered from any clinically significant toxicity experienced during treatment. Must have recovered from prior surgery or radiation. Systemic corticosteroids should be eliminated or weaned to the minimum dose before starting Ipilimumab treatment. Consult with the Medical Monitor for individual subjects
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0- 2
* Life expectancy ≥ 16 weeks
* Subjects must have the complete set of baseline (screening/baseline) radiographic images, including but not limited to brain, chest, abdomen, and pelvis. Bone scans should be completed if clinically indicated. The images can be accepted if obtained 6 weeks before initiation of Ipilimumab
* Required values for initial laboratory tests:

  1. White Blood Cells (WBC): ≥ 2000/uL (≥ 2 x 10*9*/L)
  2. Antigen Neutrophil Count (ANC): ≥ 1000/uL (≥ 1 x 10*9*/L)
  3. Platelets: ≥ 75 x 103/uL (≥ 75 x 10*9*/L)
  4. Hemoglobin: ≥ 9 g/dL (≥ 80 g/L; may be transfused)
  5. Creatinine: ≤ 2.0 x ULN
* Aspartate Aminotransferase (AST)/Alanine Aminotransferase (ALT):≤ 2.5 x Upper Limit of Normal (ULN) for subjects without liver metastasis ≤ 5 times for liver metastases
* Bilirubin: ≤ 2.0 x ULN (except for subjects with Gilbert's Syndrome, who must have a total bilirubin of less than 3.0 mg/dL)
* Men and women, at least 16 years of age
* Prior treatment with an anti-Cytotoxic T-lymphocyte Associated Protein 4 (CTLA-4) drug is allowed provided therapy was not discontinued to to drug-related toxicity
* Women of childbearing potential (WOCBP) and their partners must use highly effective methods of birth control (double barrier, e.g, condom or diaphragm or cervical cap associated with spermicide or intrauterine device combined with another form of birth control) for up to 12 weeks after the last dose of study drug to minimize the risk of pregnancy
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) at Screening and within 24 hours prior to the start of investigational product
* Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile
* Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study and for up to 12 weeks after the last dose of investigational product in such a manner that the risk of pregnancy is minimized

Exclusion Criteria:

* Women of Child-Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study and for up to 12 weeks after the last dose of investigational product
* WOCBP using a prohibited contraceptive method
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or before investigational product administration
* Subjects on any other systemic therapy for cancer, including any other experimental treatment
* Prior treatment with an anti CTLA 4 antibody if treatment failure was due to Immune-Related Adverse Events (irAEs) or discontinuation was due to an Adverse Event (AE)/Serious Adverse Event (SAE)
* Any subject enrolled in a registrational study (ie, CA184024) that has a survival endpoint should not be enrolled in CA184-045. Also, if a subject is eligible for a treatment study, he or she is not eligible for this study
* Presence of active autoimmune disease
* Presence of known hepatitis B or hepatitis C (active) infection, regardless of control on antiviral therapy
* Any subject who has a life threatening condition that requires high-dose immunosuppressants
* Subjects with melanoma who have another active, concurrent, malignant disease, with the exception of adequately treated basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* Any non-oncology vaccine therapy used for prevention of infectious diseases for up to 4 weeks before or after any dose of Ipilimumab, with the exceptions of Amantadine and Flumadine
* Any subject enrolled in a registrational study (ie, CA184-024) that has a survival as a primary endpoint should not be enrolled in CA184-045. Also, if a subject is eligible for a treatment study, he or she is not eligible for this study
* Subjects from studies CA184-042, CA184-078 or CA184-087, who are being followed for survival only or for scans only are not eligible for this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- Brazil (9):
  - Instituto do Cancer do Ceara, Fortaleza, Ceará
  - Instituto ÉTICA - AMO - Assistência Multidisciplinar em Oncologia, Salvador, Estado de Bahia
  - Instituto Nacional de Cancer - INCA, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Lucas das PUCRS, Porto Alegre, Rio Grande Do Sul (RS)
  - Hospital Mae de Deus, Porto Alegre, Rio Grande Do Sul (RS)
  - Fundacao Pio XI - Hospital De Cancer De Barretos, Barretos, São Paulo
  - Amaral Carvalho hospital, Jaú, São Paulo
  - Hospital A. C. Camargo, São Paulo, São Paulo
  - Hospital Sao Jose - Beneficencia Portuguesa - Oncology Center, São Paulo, São Paulo

REFERENCES:
- [Derived] Koguchi Y, Iwamoto N, Shimada T, Chang SC, Cha J, Curti BD, Urba WJ, Piening BD, Redmond WL. Trough levels of ipilimumab in serum as a potential biomarker of clinical outcomes for patients with advanced melanoma after treatment with ipilimumab. J Immunother Cancer. 2021 Oct;9(10):e002663. doi: 10.1136/jitc-2021-002663. PMID 34620702
- [Derived] Johnson DB, Friedman DL, Berry E, Decker I, Ye F, Zhao S, Morgans AK, Puzanov I, Sosman JA, Lovly CM. Survivorship in Immune Therapy: Assessing Chronic Immune Toxicities, Health Outcomes, and Functional Status among Long-term Ipilimumab Survivors at a Single Referral Center. Cancer Immunol Res. 2015 May;3(5):464-9. doi: 10.1158/2326-6066.CIR-14-0217. Epub 2015 Feb 3. PMID 25649350
- [Derived] Kitano S, Postow MA, Ziegler CG, Kuk D, Panageas KS, Cortez C, Rasalan T, Adamow M, Yuan J, Wong P, Altan-Bonnet G, Wolchok JD, Lesokhin AM. Computational algorithm-driven evaluation of monocytic myeloid-derived suppressor cell frequency for prediction of clinical outcomes. Cancer Immunol Res. 2014 Aug;2(8):812-21. doi: 10.1158/2326-6066.CIR-14-0013. Epub 2014 May 20. PMID 24844912
- [Derived] Iwama S, De Remigis A, Callahan MK, Slovin SF, Wolchok JD, Caturegli P. Pituitary expression of CTLA-4 mediates hypophysitis secondary to administration of CTLA-4 blocking antibody. Sci Transl Med. 2014 Apr 2;6(230):230ra45. doi: 10.1126/scitranslmed.3008002. PMID 24695685
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm